CLINICAL TRIAL: NCT06704698
Title: Paravertebral Block With Liposomal Bupivacaine and Epidural Block With Plane Bupivacaine for Postoperative Analgesia in Esophageal Surgery: A Randomized, Non-inferiority Study
Brief Title: Postoperative Analgesia Between Paravertebral Block and Epidural Block in Esophageal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, xupingbo, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2024-1037（IIT）
Record Dates: First submitted 2024-11-18; First posted 2024-11-26 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Pain Syndrome; Dizziness; Vomiting; Itching; Sweet Syndrome; Cold; Satisfaction, Patient
MeSH Terms: conditions — Somatoform Disorders; Dizziness; Vomiting; Pruritus; Sweet Syndrome; Common Cold; Patient Satisfaction | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic paravertebral block (Experimental): Ultrasound guided paravertebral block (TPVB) with liposomal bupivacaine is performed in this group. 40ml of liposomal bupivacaine and saline mixture was injected to the right T4-T5, T7-T8, and bilateral T10-T11 paravertebral spaces, with 10 ml for each space. Patient-controlled intravenous analgesia (PCIA) is used for postoperative pain management.
  Interventions: Drug: Liposomal bupivacaine
- Epidural block (Other): For the standard control group, a T6-T8 epidural block is administered. Postoperative analgesia is managed with patient-controlled epidural analgesia (PCEA).
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Liposomal bupivacaine — Thoracic paravertebral block with liposomal bupivacaine.
  Other Names: LB
  Arms: Thoracic paravertebral block
Drug: Bupivacaine Hydrochloride — Epidural block with plane bupivacaine.
  Other Names: PB (Plane Bupivacaine)
  Arms: Epidural block

SUMMARY:
Prevention of postoperative pain is essential for the recovery of esophageal surgery. Epidural analgesia is a traditional and standard perioperative pain management for these patients. Beneficials of epidural analgesia have been widely established. However, there are still several potential disadvantages such as perioperative hypotension, failure of administration, rare but serious neurological complications. Ultrasound-guided regional nerve block has become a widely used technique due to its low degree of trauma and precise target of action. In combined with liposome bupivacaine (LB), a new long-acting local anesthetic, was proven to have a maximum duration of 72 hours, thus improving postoperative analgesia, reducing opioid consumption, and enhancing patient satisfaction. The aim of this study was to evaluate the efficacy of TPVB liposomal bupivacaine (LB) or plane bupivacaine (SB) for Overall Benefit of Analgesic Score (OBAS) after esophageal surgery.

DETAILED DESCRIPTION:
After approved by the Ethics Committee of the Cancer Hospital of Zhejiang Province (Approval Number: IRB-2024-1037 (IIT)). This study was registered prior to patient admission. Written informed consent was obtained from all participants. The study is scheduled to run from November 25, 2024, to December 31, 2027. A total of 132 patients with ASA physical status I and III, undergoing thoracoscopic esophagectomy will be included. For patients in the liposomal bupivacaine group, in the left lateral decubitus position, a transversus paravertebral block (TPVB) is performed under ultrasound guidance at the right T4-T5, T7-T8, and bilateral T10-T11 paravertebral spaces, injecting 66.5mg (10 ml) liposomal bupivacaine into each space. Postoperative pain control involves patient-controlled intravenous analgesia (PCIA) with 250 μg sufentanil diluted to a total of 250 ml volume with saline. Background dose of 2-3 mL/h, PCA bolus of 2-4 mL depending on height and weight, lockout interval of 15 minutes, and a maximum dose of 10-15 mL.For the standard control group, a T6-T8 epidural block is administered, with 4-6 mL of 0.25% bupivacaine was applied depend on the height and weight. Postoperative analgesia is managed with patient-controlled epidural analgesia (PCEA), with 141 μg sufentanil and 300 mg bupivacaine hydrochloride diluted to 250 mL. Background dose of 3-6 mL/h, PCA bolus of 3-4 mL, lockout interval of 15 minutes, and a maximum dose of 20 mL.

When a participant's resting VAS score is ≥4 and they request additional pain relief, the first rescue analgesic is a single intravenous dose of acetaminophen or an NSAID (flurbiprofen axetil, 50 mg). For a second rescue, a single intravenous dose of 100 mg tramadol is administered. Additionally, the APS team adjusts the background and bolus doses based on pain relief assessments from the previous 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status I-III;
* Scheduled elective thoracoscopic esophagectomy(three-incision approach);
* Approved participation before study.

Exclusion Criteria:

* Patients with contraindications for local nerve block such as spinal anatomic structure abnormality or local infection of puncture area;
* Anergic to medications used in this study;
* Patient have chronic pain;
* Patient receiving anticoagulants, opioids or have a history of narcotic abuse or alcohol abuse;
* Inability to complete postoperative pain assessments or questionnaires due to communication barriers or mental disorders;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Benefit of Analgesic Score (OBAS) | 3 days after surgery.
  Record pain, dizziness,vomiting, itching, sweating, feeling cold, and analgesic satisfaction in the first 72 hours. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Area under the curve of mean artery pressure (MAP < 65 mmHg) | From start of anesthesia to the end of surgery, an average of 5 hours.
  Measure the area under the curve of mean artery pressure.
Visual Analog Scale (VAS) | 3 days after surgery.
  Record Visual Analog Scale scores after surgery, the scale of scores is from 0 to 10 and higher scores mean a worse outcome.
Total opioid consumption | 3 days after surgery.
  Record total opioid consumption after surgery.
In-hospital stay | From the end of surgery to discharge of hospital. An average of 10 days.
  Record in-hospital stay after surgery.

OTHER OUTCOMES:
Long time Visual Analog Scale (VAS) after surgery | 1 year.
  Record 3 months and 12 months Visual Analog Scale Scores after surgery, the scale of scores is from 0 to 10 and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangling Wang, Ph.D, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Jiangling Wang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Study plan is available when required to the principal investigator.
Supporting Information: Study Protocol
Time Frame: From the study ended to the published
Access Criteria: Doctors or healthy providers only.